CLINICAL TRIAL: NCT07389746
Title: Multimodal Prehabilitation Reduces Postoperative Complications in Highrisk Patients Undergoing Major Gastrointestinal Cancer Surgery - a Multicenter, Randomised, Controlled Trial
Brief Title: Preoperative Physical Exercise, Nutritional Support, and Psychological Preparation (Multimodal Prehabilitation) to Strengthen Patients' Overall Health and Reduce Postoperative Complications - a Multicentre Randomized, Controlled Trial
Acronym: PREHAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Cologne (Other)
Collaborators: Charity, University of Berlin (Unknown); Johannes Gutenberg University Mainz (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Robert Schier, Professor, University Hospital of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCHI1149/7-1; DFG Project#: 558914691 (Other Grant/Funding Number: German Research Society (DFG))
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cancer Surgery; Prehabilitation
Keywords: Multimodal Prehabilitation, cancer surgery, exercise, cellular mechanisms
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Multimodal Prehabilitation
  Interventions: Procedure: Multimodal Prehabilitation
- Control Group (No Intervention): Standard of Care

INTERVENTIONS:
Procedure: Multimodal Prehabilitation — Multimodal prehabilitation includes preoperative exercise (HIIT), nutritional optimization and psychological support
  Arms: Prehabilitation

SUMMARY:
In this prospective, randomized, controlled trial patients undergoing major gastrointestinal cancer surgery will be exercised (intervention group) 4 weeks before surgery with a high-intensity interval training (HIIT). They will also receive a specialized nutrition therapy and psychological support (multimodal prehabilitation). Aim of this stuy is to find out if the prehabilitation group is more resiliant to postoperative complications when compared to the control group that will receive standard of care. Another goal is to unravel the underlying mechanisms that are stimulated by exercise like enhancing vascular function, improving immune system response, strengthen cellular tumor defense and optmizing neurological outcome.

DETAILED DESCRIPTION:
Postoperative complications leading to death after surgery are the third most common cause of death (approximately one in 13 deaths). Globally this represents a significant public health challenge and is argued to be a hidden pandemic. The magnitude of this pandemic is further highlighted in a study that interrogated the American College of Surgeons NSQIP database and reported that 19% of patients had not returned home within 30 days of surgery. Additionally, the severity of postoperative complications correlates significantly with overall survival. Despite this fact, for patients presenting with advanced or recurrent gastrointestinal cancer (e.g. cancer within the pelvis; peritoneal, oesophagus, liver, stomach and pancreas) complete resection remains the only hope of survival. Approximately 85,000 Germans require major surgery for gastrointestinal cancer each year. This mandates that the reduction of postoperative complications is a high priority clinical goal.

This is the first large, multicenter prehabilitation trial (Cologne, Berlin, Tübingen and Mainz) in Germany that will integrate all aspects of modern multimodal prehabilitation to address identified modifiable preoperative risk factors in patients presenting for surgery: preoperative exercise for deconditioning, nutritional optimization, psychological intervention (these three interventions are part of our planned trial), understanding the perioperative journey and the role of the patients to be compliant with prehabilitation pathways. This contrasts other studies to date that are heterogenic and have predominantly focused on a unimodal intervention. The primary endpoint of this study => postoperative complications (Clavien-Dindo Classification grade III-V) is novel to prehabilitation studies but well-known to current large surgical multicenter trials. Our hypothesis is that prehabilitation reduces the incidence of postoperative complications and thereby has prognostic significance towards better survival.

The intended study population is a high comorbid disease cohort, with high risk of complications, increased healthcare expenditure and poor long-term cancer outcomes, as low physiological capacity and high incidence of complications are key drivers to not achieving return to intended oncological therapy.

Inclusion criteria: 1) Age ≥18/ ≤80 y; 2) Candidate for elective major abdominal cancer surgery (pelvic exenteration, cytoreductive surgery, oesophagectomy, transhiatal gastrectomy, hepatectomy, pancreatectomy, rectum resection); 3) Duke Activity Status Index score <40; 4) High risk for surgical complications defined by presence of comorbid disease as one or more of the following: 4a) Known or documented history of coronary artery disease, 4b) Known or documented history of heart failure or BNP >400pg/mL; 4c) High risk of pulmonary complications as documented by Ariscat score >4434, 4d) Diabetes currently treated with an oral hypoglycemic agent and/or insulin, 4e) Preoperative serum creatinine >200 μmol/l (>2.8 mg/dl), 4f) Morbid obesity (BMI ≥35 kg/m2), 4g) Preoperative deconditioning as confirmed by six-minute walk test (6-MWT) <400 meters or by CPET derived parameters (either anaerobic threshold (if done) <12 ml/kg/min, peak VO2 <16 mL/kg/min, peak VO2<710 mL/m2, or Ve/VCO2 [ventilator equivalents for carbon dioxide] >35); 5) Schedule allowing for at least 4 weeks for intervention with multimodal prehabilitation prior to surgery and patient's willingness to exercise Exclusion criteria: 1) Non-elective surgery; 2) Unstable cardiac or respiratory disease; 3) Locomotor limitations precluding exercise training, including severe deconditioning and frailty as reflected by inability to complete CPET test or peak VO2 <10 ml/kg/min; 4) Cognitive deterioration impeding adherence to the programme.

PREHAB intervention:

The prehabilitation programme consists of a targeted multimodal physical exercise programme and will be flanked by nutritional and psychological consultancy. Participants will be allocated to an individualized progressive preoperative exercise and education programme (intervention group) or usual care alone (control group). Participants of the control group will get written information on exercise and nutritional recommendations. General physical activity levels and nutrition behavior will be screened throughout the whole study period in both groups. Adherence to the activity program will be recorded and documented in order to conduct a per-protocol analysis.

The exercise part of the prehabilitation programme was designed by sport scientists from TU Dortmund University and the German Sport University Cologne (supervised by Prof. Zimmer and Prof. Bloch), who are experienced in implementing and conducting comparable programmes for various clinical populations, including cancer patients (e.g. a recent H2020 exercise trial with breast cancer patients, https://www.h2020preferable.eu/partners/). Within the preparation phase (months 1-6), teaching and documentation material for the exercise programme as well as an 'Exercise SOP' will be prepared and delivered to all study centres. All study sites will conduct the same exercise programme in accordance with the exercise SOP. Regular video meetings of sports therapists of each site with the responsible sports scientists from TU Dortmund University and the German Sport University Cologne will be conducted weekly in order to keep track of intervention fidelity and Borg scale consistency.

The overall aim of this programme is to maximize the physical capacity (in regards of strength and endurance) within the given time frame. The supervised progressive exercise programme will be conducted and supervised by a professional sport therapist, consisting of three 50-min sessions per week. Each session will be divided in (i) a resistance exercise part, aiming to increase patients' strength and (ii) an endurance part aiming to improve patients' cardio-respiratory fitness. A home-based walking programme (as per usual care) will be conducted in the intervention group on the days, when they are not attending the prehabilitation programme.

Progressive Resistance Training (20 min) Three different machine-based exercises for major muscle groups (Squat, Bench press, Rowing) Three sets, 10-12 repetitions, with 90 seconds recreational breaks Weights will be progressively and individually adjusted to self- perceived exhaustion (RPE-Scale) so that patients will be able to complete a minimum of eight and maximum of twelve repetitions. Initial load will be adjusted based on validated 12-RM assessment.

Progressive Endurance Training (30 min)

Cycle-based periodised ergometer training, consisting of moderate continuous training (MCT) and high-intensity interval training (HIIT). Periodization between sessions:

First week: MCT - MCT - MCT Second week: MCT - HIIT - MCT Third week: HIIT - MCT - HIIT Fourth week: HIIT - HIIT - HIIT Intensity will be adjusted according to peak power output (PPO) reached at the initial CPET.

MCT: 5 min warm-up, 20 min continuous at 60% PPO, 5 min cool-down HIIT: 5 min warm-up, 5 intervals for 1.5 min at 85-90% PPO with 3 min unloaded pedalling between intervals, 5 min cool-down.

Deep breathing exercise / Spirometer

The prehabilitation group will perform deep breathing exercise (DBE) training with incentive spirometer (IS) under supervision at the first prehabilitation visit and at home daily twice (morning & evening) over 4 weeks preoperatively. IS training instructions will be given practically by the sports medicine staff before the first exercise session. The experts will first introduce the IS and explained how it is used with a demonstration of the proper position how to hold the IS during the exercise. The steps of inspiration, holding the breath in and expiration will be performed under supervision. The DBE session will take 20 minutes, containing of the following protocol and instruction to the patient: 1) Position: Sitting upright in a chair or bed, 2) Setup: Instruction to exhale normally, then place the mouthpiece in mouth, sealing lips tightly, 3) Inhaling: Breathing in slowly and deeply through mouth, watching the piston or ball of the spirometer rise, 4) Target: Aim for the indicator to stay between the arrows or reach your set goal (if marked), 5) Instruction not to breathing too fast as it makes the ball shoot up and not too slow as it stays low, 6) Holding phase: Patient holds breath at the top for 3 to 5 seconds, 7) Exhalation phase: Patient removes the mouthpiece and exhales normally, 8) Cough: Patient is instructed to give a deep, strong cough to clear mucus, 9) Rest & Repeat: Patient rests briefly and repeats up to 5 times over 20 minutes.

Nutritional Intervention In the preoperative phase (5 weeks before surgery => see trial visits table), a registered dietitian will perform an initial assessment on nutritional and dietary habits in the intervention group with the modified Patient-generated subjective global assessment (PG-SGA SF)36,37 and the Malnutrition Universal Screening Tool (MUST)38,39. Also, a 3-day total food diary will be conducted by the intervention group to evaluate the individual risk of malnutrition (one or more of the following: PG SGA SF≥4, MUST≥2, BMI<20, Serum albumin <30 g/L). Based on the results of the assessment above, nutritional intervention will be performed by an ecotrophologically-trained physician and/or a clinician assistant (dietician) by designing an individual nutrition care plan on appropriate food choices and fluid intake to meet their nutritional needs with considerations of optimal meal size, supplements (protein supplement) and increased nutrient density. Whey protein supplement will be prescribed to guarantee a daily protein intake of min. 1.5 g/kg of current body weight. These supplements will be consumed immediately after exercise during training days or every morning after breakfast. In cases with risk of vitamin deficiencies (e.g. Vitamin D), vitamin supplementation according to the 3-day total food diary will be advised. Additionally, all participants regardless to their individual risk of malnutrition receive intensive counselling in order to optimize eating habits (e.g. higher intake of vegetables and fruits, recommendations regarding life style risks and a stop smoking / alcohol drinking program will be offered). Once a week the patients will be contacted by phone to support and re-evaluate the individual nutritional concepts by ecotrophologically-trained physician and/or a clinician assistant (dietician).

Psychological Intervention The psychological intervention aims at decreasing distress and increasing emotional wellbeing. The psychological intervention will be conducted in the preoperative phase (4 weeks until 2 days before surgery => see trial visits table) either in person at the study centres or via video, depending on the patients' preference. We will statistically control the method of implementation (face-to-face or video) in subgroup analyses. Each psychological intervention lasts 30 (+/- 5) minutes. A clinician assistant (CA) trained in the appropriate techniques will carry out the psychological intervention in a 1-to-1 session. In the first session, the CA introduces him / herself and explains the content and aim of the psychological intervention. Every session starts with 10 minutes of Progressive Muscle Relaxation (PMR) according to Jacobsen. The CA then discusses the exercise with the patient (e.g. feasibility, exercise experience, differences in perception of tension and relaxation). Afterwards, the patient is instructed in a deep breathing exercise. The CA hands out a CD with instructions on relaxation techniques to the patient and encourages her/ him to use relaxation techniques twice a day (e.g. in the morning and evening) over the following weeks. If there is still time after these two exercises, the CA will involve the patient in a talk about his/ her psychological resources (i.e. family and friends, pets, hobbies, interests) or themes considered as pleasant by the patient. At the beginning of sessions 2, 3 and 4, the CA will politely ask the patients whether she/ he has had the opportunity to use the relaxation techniques in the last week and document the patients' answers. This serves on the one hand to increase patient adherence to regularly perform relaxation techniques, but also to be able to draw cautious conclusions about patient's adherence to regularly performing relaxation techniques. We will assess the level of mental distress using the Generalized Anxiety Disorder 7 (GAD-7) Questionnaire before and after the 4 weeks' prehabilitation programme as well as postoperatively on days 1, 3, 5 and / or day of discharge. If an increased level of distress is detected by the GAD-7 (GAD-7 score >= 10), patients will be referred to a professional clinical psychologist as part of an in-hospital council.

Outcome measures

Outcome measures will be assessed by a blinded study endpoint committee of two independent researchers. Inter-observer variability will be analysed and reported.

Primary endpoint: Postoperative complications (Clavien-Dindo-Classification grade III-V). This is a well-known, metric and validated outcome parameter that is sensitive to surgical risk and prognostic association to long-term (five-year) survival in cancer patients. We will analyse this outcome in the context of clinically relevant time window (30days after surgery or time of patient's discharge), where, based on our preliminary data, most of the CDIII-V complications occur.

Preliminary prehabilitation studies have shown that it is feasible to exercise patients preoperatively and improve functional capacity. Further RCTs have been conducted recently adding to the body of evidence that prehabilitation has beneficial effects in reducing complications. However, these studies mainly consider colorectal and not upper gastrointestinal cancer patients as in our planned trial. This group of patients is facing rather high complication risk of 30-40%.

Secondary endpoints: 1) Postoperative Comprehensive Complication Index (CCI), 2) Medical complications (i.e. cardiac, pulmonary, sepsis => all complications will be predefined in protocol); 3) Length of ICU stay (LOICUS), Hospital Length of Stay (HLOS), Days at home after surgery (DAH-30)4, time / number of patients to start postoperative adjuvant therapy 4) Cost-effectiveness / -utility analysis (RAND, iPCQ/iMCQ); 5) Functional capacity (CPET, DASI); 6) Quality of life (HRQoL, EORTC QLQ-C30), incidence of perioperative anxiety disorder / depression (GAD-7)

7) Biobanking: In addition to all endpoints mentioned above, serum / peripheral blood mononuclear cells (PBMCs) and tumour material will be stored for mechanistic analysis (e.g. inflammation, wound healing, immune function) in secondary step. Putative biological mechanisms attributed to the effectiveness of prehabilitation include the pleiotropic effects of exercise, which through numerous physiological systems may impact surgical outcome. Exercise as part of prehabilitation stimulates bone-marrow derived cells improving vascular function and wound healing. An episode of maximal exercise mobilised progenitor populations into the peripheral circulation in some patients and this was associated with fewer postoperative complications. Exercise also generates erythropoietin, increasing red cell counts and stimulates natural killer cell production, which may modulate the tumour defence response. Recent evidence suggests that preoperative exercise may down-stage tumour grade. These beneficial effects may be driven by exercise-induced anti-inflammatory pathways as well as by a mobilisation and activation of tumour-competitive lymphocytes. The above mechanisms will be investigated in consecutive analyses with regard to the research topics: 1. endothelial regeneration, 2. inflammation 3. tumour defense and 4. cognitive function. An additional research proposal ("Sachbehilfeantrag") will be submitted in order to clarify on the specific translational mechanisms (i.e. exercise-stimulation of natural killer cells for clinical tumour defense) and to apply for additional funding for the analyses. An additional research proposal ("Sachbeihilfeantrag") will be submitted in order to clarify on the specific translational mechanisms and to apply for additional funding for the analyses.

Methods against bias

Subject enrolment is consecutive (i.e. no convenience sample). Selection bias is minimized by random assignment with ratio 1:1 stratified by tumour entity as followed:

1. Upper GI => oesophagectomy, transhiatal gastrectomy
2. Lower GI => pelvic exenteration, cytoreductive surgery, rectum resection
3. Hepato-Pancreato-Biliary surgery (HPB) => hepactectomy, pancreatectomy

The randomization procedure is based on permuted blocks of varying length and implemented as a central 24/7 Internet service (i.e. ALEA, FormsVision BV, Abcoude, NL). Performance bias is minimized by carefully following the study protocol and continuous monitoring of adherence. Single-blinding of the statistician analyzing the data will be performed. Attrition bias is minimized by provision of excellent and free medical care and subject management by dedicated trained study personnel. Detection bias is minimized by careful standardization and masking of outcome assessment as far as possible. The measurement of key outcome measures (complication, LOICUS, HLOS, DAH-30) is at low risk of bias.

Proposed sample size / power calculations

We assume a percentage of patients with at least one Clavien-Dindo grade III postoperative complication of 35% in the control group (CON) (based on the literature and own pilot data/ see Table 3) and a 40% relative reduction based on the experimental prehabilitation intervention (EXP), thus an absolute reduction of 14% points to 21% (EXP). This seems a cautionary assumption since Barberan-Garcia et al.48 report a relative reduction of 50%. Assuming 80% power at two-sided significance level 5%, Pearson's chi-squared test requires n=161 subjects per group, i.e., n=322 subjects in total (Stata/SE 16.1, StataCorp LLC, College Station, TX, USA). Further assuming 20% attrition (e.g., due to inadherence, discontinuation of prehabilitation, loss to follow up) n=403 (≈322/0.8) subjects need to be enrolled and randomised in total (to be analysed according to the intention-to-treat). We assume that cluster effects due to therapist or physician are neglectable for power calculation, however they will be explored in the statistical analysis.

Compliance / rate of loss to follow-up

We expect patients to welcome the cost-free exercise testing before their surgery in order to find out at what physiological capacity level they start their perioperative course. The interventional group receives an individually tailored exercise plan, that is motivating and less time consuming. Further, the type of exercise programme (interval training) is patient friendly and will be adapted to their physical capability. Nevertheless, we anticipate a 20% drop-out rate of our study cohort (e.g., due to inadherence, discontinuation of prehabilitation) and adjusted our sample size accordingly.

8.10 Feasibility of recruitment / access to study population

Being large University Hospitals, the four included study sites (Cologne, Berlin, Mainz and Tübingen) perform a sufficient number of surgeries (250-300 major abdominal surgery cases per year per study site) in order to recruit enough patients for the proposed sample size (n= 403). Furthermore, a sufficient number of postoperative complications is anticipated in our study cohort justified on the basis of clinical data (n=663, 2016-2020) for oesophagectomy patients at the University Hospital of Cologne. Taking into account that it is a high-volume centre with high expertise, still 50% of the esophagectomy patients suffered a complication Clavien-Dindo ≥III.

Summarized below are the included surgery types and their representative complication rates as described in the literature. High surgical aggression (50% complication rate): i.e. oesophagectomy, pancreaticoduodenectomy, transhiatal gastrectomy. Intermediate surgical aggression (30% complication rate): i.e. gastric bypass, total colectomy, rectal resection, major liver resection, pancreas resection. Minor surgical aggression (10% complication rate): partial gastrectomy, sleeve gastrectomy, segmental colon resection, minor liver resection, Clavien-Dindo complications grade III-V are described within 10% after liver resection and 38% after pancreatectomy, therefore quite a number of grade III-V complications can be expected in our study cohort in order to ensure the feasibility of our study endpoint. We know from previous studies that the type of preoperative exercise that will be conducted in this trial is entertaining and adequately adopted to the patient's physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* Candidate to elective major gastrointestinal cancer surgery (pelvic exenteration, cytoreductive surgery, oesophagectomy, transhiatal gastrectomy, hepatectomy, pancreatectomy, rectum resection)
* High risk for surgical complications defined by presence of comorbid disease such as deconditioning, heart disease, diabetes, renal impairment or morbid obesity
* Duke Activity Status Index score (DASI) <402
* Schedule allowing for at least 4 weeks for intervention with multimodal prehabilitation prior to surgery / willingness to exercise

Exclusion Criteria:

* Non-elective surgery
* Unstable cardiac or respiratory disease
* Locomotor limitations precluding exercise training
* Cognitive deterioration impeding adherence to the programme
* Enrolment in other research studies affecting study endpoint

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications defined as Clavien-Dindo Classification grade III-V | Postoperative complications (Clavien-Dindo Classification grade III-V) is a well-known, metric and validated outcome parameter that is sensitive to surgical risk and prognostic association to long-term (five-year) survival in cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No
Not permitted by ethical protocol